CLINICAL TRIAL: NCT02536131
Title: Intestinal Microbiome and Psychological Correlates in Irritable Bowel Syndrome and Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gabriele Moser, Prof. Dr. Gabriele Moser, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EK 1502/2014
Record Dates: First submitted 2015-08-21; First posted 2015-08-31 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: IBS; IBD
Keywords: Psychosomatics; Gastroenterology; Psychoneuroimmunology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study group (Other): 7-10 sessions gut-directed hypnotherapy within 12 weeks
  Interventions: Other: Gut-directed hypnotherapy

INTERVENTIONS:
Other: Gut-directed hypnotherapy — relaxation technique with hypnotic induction and suggestions aimed at fostering sense of control, acceptance and calming of bowels.
  Other Names: Gut-focused hypnotherapy

SUMMARY:
Longitudinal Investigation of intestinal microbiome, fecal inflammation markers, stress and psychological variables in patients with irritable bowel syndrome and inflammatory bowel disease undergoing gut-directed hypnotherapy (GHT).

DETAILED DESCRIPTION:
Study design is a within-subject design with assessment at 4 points in time. Data will be collected 3-1 month before first GHT session (T1), immediately before first session (T2), at the last session (T3), and 3-6 months after last session (T4).

Study patients will be recruited consecutively at the special outpatient-clinic for psychosomatics at the division of Gastroenterology and Hepatology, department for Internal Medicine III, University Hospital Vienna.

Patients undergo GHT in group setting, which has been shown to reduce irritable bowel syndrome (IBS) symptoms and to increase psychological wellbeing. The GHT protocol used will be the Manchester protocol of gut-directed hypnotherapy and consists of 10 weekly sessions (45 minutes) with six up to eight patients per group over a treatment period of 12 weeks.

The following variables will be assessed using standardized questionnaires: anxiety and depression (HADS-D), perceived stress (PSQ), resilience (CDRISC), and quality of life (visual analogue scales). IBS symptoms will be captured by the IBS Severity Scoring System (IBS-SSS), inflammatory bowel disease (IBD) disease activity via Harvey-Bradshaw-Index. Additionally, medication intake and food supplements will be assessed.

Microbiome data will be gained by frozen stool samples, collected by patients at home. Patients will be provided with a delivery kit to keep the samples frozen. Patients are asked to collect the first stool of the day and not to change diet, medication and intake of pre/probiotics during the hole study period, if possible (documented). At each time point (T1-T4) patients are ask to bring two immediately frozen (stored in their home freezer) double samples (2 stool samples within 1 week) to the hospital to be immediately stored at minus 20 degree Celsius. If patients do not have a home freezer, stool will be collected and frozen at the hospital.

Planned analyses comprise longitudinal and cross-sectional comparisons Intestinal colonization will enter in the analyses according to an algorithm assigning values for an increase or reduction of dysbiosis. Dysbiosis is hereby defined by the following markers: reduction of fecal biodiversity, lowered occurrence of the species Bifidobacterium, Lactobacillus and Faecalibacterium prausnitzi, increased occurrence of Enterobacteriaceae, and a higher quotient Firmicutes:Bacteroidetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBS or IBD
* Eligible for gut-directed hypnotherapy
* Adult age (18-89)
* Sufficient knowledge of german language

Exclusion Criteria:

* Severe somatic or psychiatric illness
* Operations of the GI tract

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Changes in gut microbiome as assessed through analyzing fecal samples | 7 days
  Analysis of faeces by taxonomic and functional classification via 16s ribosomal ribonucleic acid (rRNA) sequencing with special regard to commensal microbiota and pathobionts
Perceived Stress Questionnaire | 10 days
Hospital Anxiety and Depression Scale | 7 days
  Total score as a measure of psychological distress

SECONDARY OUTCOMES:
Connor-Davidson Resilience Scale | 10 days
Severity Scoring System for Irritable Bowel Syndrome | 10 days
Faecal calprotectin | 1 day
  Intestinal inflammation marker
Harvey-Bradshaw-Index | 2 days
  Disease activity index for IBD's
Quality of life visual analogue scales | 10 days
  Visual analogue scales pertaining to physical, psychological and general wellbeing
GI single symptom visual analogue scales | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Moser, MD, Prof, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Peter J, Fournier C, Durdevic M, Knoblich L, Keip B, Dejaco C, Trauner M, Moser G. A Microbial Signature of Psychological Distress in Irritable Bowel Syndrome. Psychosom Med. 2018 Oct;80(8):698-709. doi: 10.1097/PSY.0000000000000630. PMID 30095672